CLINICAL TRIAL: NCT01292915
Title: Survey of Non-Variceal Upper Gastro Intestinal Bleeding in Vietnamese Patients
Acronym: NIS-PUB
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GVN-DUM-2010/1
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Re-bleeding in NVUGIB
Keywords: Re-bleeding, NVUGIB

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The main aim of the study is to describes the outcomes of patients with Upper Gastrointestinal Bleed (UGIB) in a real-life setting. Additionally analyse assessed predictors of outcome, including the impact of hemostatic endoscopic and pharmacologic therapies.

DETAILED DESCRIPTION:
MSD

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>=18yrs) admitted to the hospital, or inpatients admitted for another reason, presenting with overt non-variceal upper GI bleed manifesting as hematemesis/coffee ground vomiting, melena, hematochezia...
* Evidence that an upper GI endoscopy was performed

Exclusion Criteria:

* GI bleeding not from NVUGIB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NVUGIB patients in 13 hospitals in Hanoi, HCMC, Danang
Sampling Method: Non-Probability Sample
Enrollment: 1044 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Rebleeding (within 7 days from the Non-Variceal Upper Gastro Intestinal Bleeding (NVUGIB) episode) | 7 days

SECONDARY OUTCOMES:
Surgery due to re-bleeding | 7 days
Mortality due to bleeding | 7 days
Rebleeding in high risk peptic ulcer patients | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Dao Van Long, MD,PhD, Principal Investigator — Hanoi Medical University
Locations (3):
- Vietnam (3):
  - Research Site, Da Nang
  - Research Site, Hanoi
  - Research Site, HoChiMinh City

REFERENCES:
- See also: CSR_Synopsis_NIS-GVN-DUM-2010_1 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=894&filename=CSR_Synopsis_NIS-GVN-DUM-2010_1.pdf